CLINICAL TRIAL: NCT01119378
Title: Calcium Absorption Efficiency As An Indicator For Vitamin D Sufficiency
Brief Title: Study to Observe the Capability to Absorb Calcium as an Measure of Adequate Levels of Vitamin D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Principal Investigator, John F. Aloia, MD, Principal Investigator, Winthrop University Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 10003
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Postmenopausal; Vitamin D Deficiency
Keywords: Post menopausal; Vitamin D sufficiency; Calcium absorption efficiency; Dual isotope technique
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Post Menopausal (Experimental): post menopausal women between the ages 50-70 yrs.
  Interventions: Other: Dual isotope technique

INTERVENTIONS:
Other: Dual isotope technique — Dual isotope technique using stable isotopes
  Other Names: Kinetic study; dual stable isotope

SUMMARY:
The purpose of this study is to determine the capability to absorb calcium as a measure of the sufficient levels of Vitamin D. Calcium absorption will be measured at baseline and after vitamin D3, by dual calcium isotope technique using stable isotopes in post menopausal women between the ages 50 and 70yrs. Subjects will have a screening visit, first and final visits. Subjects will be randomly assigned to a placebo or daily doses of vitamin D3. The specific aim of this study is to determine the level of vitamin D that will maximize the absorption of calcium and establish the relationship between the administered calcium dose and the actual absorbed calcium dose versus administered dose of Vitamin D and the serum levels of Vitamin D.

DETAILED DESCRIPTION:
The specific aims of this project are:

1. To determine the level of 25OHD that maximizes calcium absorption efficiency.
2. To describe the dose response curve of calcium absorption to vitamin D intake and serum 25OHD.

This will be a randomized, double-blind, placebo-controlled trial of healthy postmenopausal females to determine the individual and combined effects of calcium and vitamin D supplementation.70 female participants, ages 50 to 70 years of age who are menopausal for over 1 year will be recruited into the study . The patients participation in this study will last about 10 weeks. Approximately 70 subjects from Winthrop University Hospital and the surrounding area will participate in this study. There is a total of 3 visits. Patients will be fasting for all visits. The first visit is a screening visit to determine if the patients qualify.

At visit 2, the patients will be given a light breakfast and asked to drink an 8 ounce glass of milk or calcium fortified orange juice containing a calcium isotope. After breakfast, the doctor or nurse will start an intravenous infusion and inject the patient with an IV solution containing a calcium isotope. This is a stable calcium isotope that is not radioactive and has no known toxicity. The patients will also be asked to collect a 24 hour urine and return it to us the next day.

The volunteers will be divided into four groups:

The first group will take 800 iu daily of vitamin D supplementation. The second group will take 2000 iu daily of vitamin D.The third group will take 4000 iu vitamin D and the fourth group will only take placebos. Visit 3 is essentially the same as visit 2, with subjects returning unused study medication and given new tablets

Food frequency questionnaires will be filled out at the initial visit and final visit. Diet will be assessed using 3-day diet history form and NutritionPro analysis software. Patients will be asked to refrain from taking other vitamin D supplements and to continue their usual calcium intake.

ELIGIBILITY:
Inclusion Criteria:

Post menopausal women between the ages 50-70 yrs.

Exclusion Criteria:

1. Any chronic medical illness including diabetes mellitus, history of myocardial infarction, or heart failure, malignancy, uncontrolled hypertension, history of anemia, leukemia, or other hematologic abnormalities, lupus, rheumatoid arthritis, or other rheumatologic disease, or kidney disease of any kind as determined by history and physical examination.
2. Subjects with a BMI >35kg/m2
3. Use of medication that influences vitamin D and bone metabolism (i.e. anticonvulsant medications, glucocorticoids, HAART [AIDS treatment], antirejection medications, high dose diuretics etc).
4. Significant deviation from normal either in history, physical examination, or laboratory tests as evaluated by the primary investigator.
5. Patients with a history of hypercalciuria ( Urine calcium:creatinine ratio > 0.37 , hypercalcemia ( serum calcium >10.21, nephrolithiasis, and active sarcoidosis will also be excluded.
6. Unexplained weight loss >15% during the previous year or history of anorexia nervosa
7. Participation in another investigational trial in the past 30 days prior to the screening evaluation.
8. Patients reporting alcohol intake greater than 2 drinks daily.
9. Subjects with baseline 25-OHD level greater than 70 nmol /L will be excluded.
10. Smokers greater than one pack per day will be excluded
11. Dietary calcium intake greater than 2000 mg will be excluded
12. Participants who have history of allergy to milk, gluten or orange juice will be excluded
13. Participants willing not to forego multivitamins and vitamin D supplements during the study -

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To determine the level of 25OHD that maximizes calcium absorption efficiency. | 3 months

SECONDARY OUTCOMES:
To describe the dose response curve of calcium absorption to vitamin D intake and serum 25OHD | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: John F Aloia, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States

REFERENCES:
- [Derived] Aloia JF, Dhaliwal R, Shieh A, Mikhail M, Fazzari M, Ragolia L, Abrams SA. Vitamin D supplementation increases calcium absorption without a threshold effect. Am J Clin Nutr. 2014 Mar;99(3):624-31. doi: 10.3945/ajcn.113.067199. Epub 2013 Dec 11. PMID 24335055